CLINICAL TRIAL: NCT01706783
Title: A Randomised, Open-labelled, Active-controlled, Multiple Dose, Dose Escalating, Sequential Dose Group Trial Investigating Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Once-weekly Long-acting Growth Hormone (NNC0195-0092, Somapacitan) Compared to Once-daily Norditropin NordiFlex® in Adults With Growth Hormone Deficiency
Brief Title: A Trial Investigating the Safety, Tolerability, Availability and Distribution in the Body of Once-weekly Long-acting Growth Hormone (Somapacitan) Compared to Once Daily Norditropin NordiFlex® in Adults With Growth Hormone Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN8640-3947; 2011-005484-24 (EudraCT Number); U1111-1125-7331 (Other: WHO)
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — somapacitan; NNC0195-0092; Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC0195-0092 (somapacitan) (Experimental)
  Interventions: Drug: somapacitan
- Norditropin NordiFlex® (Active Comparator)
  Interventions: Drug: Norditropin NordiFlex®

INTERVENTIONS:
Drug: somapacitan — Subcutaneous (s.c., under the skin) administration once weekly (Days 1, 8, 15 and 22) of 4 different doses of NNC0195-0092 (somapacitan) in an escalating order
  Other Names: NNC0195-0092
  Arms: NNC0195-0092 (somapacitan)
Drug: Norditropin NordiFlex® — Subcutaneous (s.c., under the skin) administration daily for 28 days. The daily dosing will be the same as the pre-trial daily dose of human growth hormone (hGH) taken by the adult with growth hormone deficiency
  Arms: Norditropin NordiFlex®

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the safety, tolerability, availability and distribution in the body of once-weekly long-acting growth hormone (NNC0195-0092, somapacitan) compared to once daily Norditropin NordiFlex® in adults with growth hormone deficiency (GHD).

ELIGIBILITY:
Inclusion Criteria:

* Adults with GHD as defined in the consensus guidelines for the diagnosis and treatment of adults with GHD
* Stable human growth hormone (hGH) replacement therapy for at least 3 months

Exclusion Criteria:

* Participation in another clinical trial within 3 months or receipt of any investigational medicinal product within 3 months prior to randomisation
* Active malignant disease or malignant disease within the last 5 years with exception of fully treated local basal cell carcinoma or carcinoma in situ of cervix
* Proliferative retinopathy judged by retina-photo within the last year - only with concomitant diabetes
* Heart insufficiency, New York Heart Association (NYHA) class above 2
* Adults with GHD with poorly controlled diabetes mellitus with a glycosylated haemoglobin (HbA1c) 64 mmol/mol (8.0%) and/or insulin treatment
* Stable pituitary replacement therapy for less than 3 months

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-10-12 (Actual); Primary Completion 2013-11-18 (Actual); Study Completion 2013-11-18 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | From first administration of trial product and up until Day 49

SECONDARY OUTCOMES:
NNC0195-0092 (somapacitan) only: Area under the curve, AUC (0-168h) | From 0 to 168 hours
Norditropin NordiFlex® only: AUC (0-24h) | From 0 to 24 hours
NNC0195-0092 (somapacitan), first dose administration only: AUC (0-168h) | From 0 to 168 hours
Norditropin NordiFlex®, first dose administration only: AUC (0-24h) | From 0 to 24 hours
NNC0195-0092 (somapacitan): Maximum serum concentration (Cmax) | From 0 to 168 hours
Norditropin NordiFlex®: Cmax | From 0 to 24 hours
Insulin-like growth factor I (IGF-I): AUC (0-168h) | From 0 to 168 hours
IGF-I: Cmax | From 0 to 168 hours
Insulin-like growth factor binding protein-3 (IGFBP-3): AUC IGFBP-3(0-168h) | From 0 to 168 hours
IGFBP-3: Cmax | From 0 to 168 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (4):
- Denmark (3):
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, København Ø
  - Novo Nordisk Investigational Site, Odense
- Novo Nordisk Investigational Site, Stockholm, Sweden

REFERENCES:
- [Background] Juul Kildemoes R, Hojby Rasmussen M, Agerso H, Overgaard RV. Optimal Monitoring of Weekly IGF-I Levels During Growth Hormone Therapy With Once-Weekly Somapacitan. J Clin Endocrinol Metab. 2021 Jan 23;106(2):567-576. doi: 10.1210/clinem/dgaa775. PMID 33313798
- [Derived] Papathanasiou T, Agerso H, Damholt BB, Hojby Rasmussen M, Kildemoes RJ. Population Pharmacokinetics and Pharmacodynamics of Once-Daily Growth Hormone Norditropin(R) in Children and Adults. Clin Pharmacokinet. 2021 Sep;60(9):1217-1226. doi: 10.1007/s40262-021-01011-3. Epub 2021 Apr 17. PMID 33864240
- [Derived] Juul RV, Rasmussen MH, Agerso H, Overgaard RV. Pharmacokinetics and Pharmacodynamics of Once-Weekly Somapacitan in Children and Adults: Supporting Dosing Rationales with a Model-Based Analysis of Three Phase I Trials. Clin Pharmacokinet. 2019 Jan;58(1):63-75. doi: 10.1007/s40262-018-0662-5. PMID 29671202
- [Derived] Rasmussen MH, Janukonyte J, Klose M, Marina D, Tanvig M, Nielsen LF, Hoybye C, Andersen M, Feldt-Rasmussen U, Christiansen JS. Reversible Albumin-Binding GH Possesses a Potential Once-Weekly Treatment Profile in Adult Growth Hormone Deficiency. J Clin Endocrinol Metab. 2016 Mar;101(3):988-98. doi: 10.1210/jc.2015-1991. Epub 2016 Jan 4. PMID 26727076
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com